CLINICAL TRIAL: NCT04487080
Title: A Phase 3, Randomized Study of Amivantamab and Lazertinib Combination Therapy Versus Osimertinib Versus Lazertinib as First-Line Treatment in Patients With EGFR-Mutated Locally Advanced or Metastatic Non-Small Cell Lung Cancer.
Brief Title: A Study of Amivantamab and Lazertinib Combination Therapy Versus Osimertinib in Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Acronym: MARIPOSA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR108856; 73841937NSC3003 (Other: Janssen Research & Development, LLC); 2020-000743-31 (EudraCT Number); 2023-506576-27-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2020-07-23; First posted 2020-07-27 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — amivantamab; osimertinib; lazertinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only Arm B and C will be masked to all (Double-blind).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment Arm A (Open-label): Amivantamab and Lazertinib (Experimental): Participants will receive amivantamab 1050 milligram (mg) intravenously (IV) for body weight less than (<) 80 kilogram (kg) and 1400 mg for body weight greater than or equal to (>=) 80 kg in 28-day cycles: once weekly in Cycle 1 (with a split dose on Days 1-2), and then every 2 weeks in subsequent cycles. Lazertinib will be administered 240 mg (80*3) orally once daily.
  Interventions: Drug: Amivantamab; Drug: Lazertinib
- Treatment Arm B (Double-blind): Osimertinib+Placebo Lazertinib (Active Comparator): Participants will receive osimertinib 80 mg orally once daily plus matching placebo of lazertinib 240 mg (80*3) orally once daily.
  Interventions: Drug: Osimertinib; Drug: Placebo
- Treatment Arm C (Double-blind): Lazertinib+Placebo Osimertinib (Experimental): Participants will receive lazertinib 240 mg (80*3) orally once daily plus matching placebo of osimertinib 80 mg orally once daily.
  Interventions: Drug: Lazertinib; Drug: Placebo

INTERVENTIONS:
Drug: Amivantamab — Participants will receive amivantamab intravenously.
  Other Names: JNJ-61186372
  Arms: Treatment Arm A (Open-label): Amivantamab and Lazertinib
Drug: Osimertinib — Participants will receive osimertinib capsules orally.
  Arms: Treatment Arm B (Double-blind): Osimertinib+Placebo Lazertinib
Drug: Lazertinib — Participants will receive lazertinib tablets orally.
  Other Names: JNJ-73841937 and YH-25448
  Arms: Treatment Arm A (Open-label): Amivantamab and Lazertinib; Treatment Arm C (Double-blind): Lazertinib+Placebo Osimertinib
Drug: Placebo — Participants will receive matching placebo orally.
  Arms: Treatment Arm B (Double-blind): Osimertinib+Placebo Lazertinib; Treatment Arm C (Double-blind): Lazertinib+Placebo Osimertinib

SUMMARY:
The purpose of this study is to assess the efficacy of the amivantamab and lazertinib combination, compared with osimertinib, in participants with epidermal growth factor receptor (EGFR) mutation (Exon 19 deletions [Exon 19del] or Exon 21 L858R substitution) positive, locally advanced or metastatic non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Participant must have newly diagnosed histologically or cytologically confirmed, locally advanced or metastatic non-small cell lung cancer (NSCLC) that is treatment naive and not amenable to curative therapy including surgical resection or chemoradiation
* The tumor harbors exon 19 deletions (Exon 19del) or Exon 21 L858R substitution, as detected by an food and drug administration (FDA)-approved or other validated test in a clinical laboratory improvement amendments (CLIA) certified laboratory (sites in the United states [US]) or an accredited local laboratory (sites outside of the US) in accordance with site standard of care
* Mandatory submission of unstained tissue from tumor (in a quantity sufficient to allow for central analysis of EGFR mutation status and blood (for circulating tumor deoxyribonucleic acid [ctDNA], digital droplet polymerase chain reaction [ddPCR], and pharmacogenomic analysis)
* Any toxicities from prior anticancer therapy must have resolved to common terminology criteria for adverse events (CTCAE) Grade 1 or baseline level
* Participant must have at least 1 measurable lesion, according to response evaluation criteria in solid tumors (RECIST) v1.1 that has not been previously irradiated. Measurable lesions should not have been biopsied during screening, but if only 1 non-irradiated measurable lesion exists, it may undergo a diagnostic biopsy and be acceptable as a target lesion, provided the baseline tumor assessment scans are performed at least 14 days after the biopsy

Exclusion Criteria:

* Participant has received any prior systemic treatment at any time for locally advanced Stage III or metastatic Stage IV disease (adjuvant or neoadjuvant therapy for Stage I or II disease is allowed, if administered more than 12 months prior to the development of locally advanced or metastatic disease)
* Participant has an active or past medical history of leptomeningeal disease
* Participant with untreated spinal cord compression. A participant that has been definitively treated with surgery or radiation and has a stable neurological status for at least 2 weeks prior to randomization is eligible provided they are off corticosteroid treatment or receiving low-dose corticosteroid treatment less than or equal to (<=) 10 milligrams per day (mg/day) prednisone or equivalent
* Participant has an active or past medical history of interstitial lung disease (ILD)/pneumonitis, including drug-induced or radiation ILD/pneumonitis
* Participant has known allergy, hypersensitivity, or intolerance to the excipients used in formulation of amivantamab, lazertinib, or osimertinib, or any contraindication to the use of osimertinib
* Participant has symptomatic brain metastases. A participant with asymptomatic or previously treated and stable brain metastases may participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1074 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2027-06-29 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (267):
- United States (20):
  - Arizona Oncology Associates, PC - HAL, Goodyear, Arizona
  - Yuma Regional Medical Center, Yuma, Arizona
  - City of Hope Long Beach Elm, Long Beach, California
  - University of California Irvine, Orange, California
  - Rocky Mountain Cancer Centers, Lone Tree, Colorado
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - University Cancer And Blood Center LLC, Athens, Georgia
  - East Jefferson General Hospital, Metairie, Louisiana
  - Maryland Oncology Hematology, PA, Columbia, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Minnesota Oncology Hematology P A, Edina, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School Of Medicine, St Louis, Missouri
  - Astera Cancer Care, East Brunswick, New Jersey
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology P A, Austin, Texas
  - Oncology Consultants Texas, Houston, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
- Argentina (5):
  - Centro Oncológico Korben, Buenos Aires
  - Instituto Alexander Fleming, Buenos Aires
  - Hospital Privado Centro Medico de Cordoba, Córdoba
  - Centro Oncologico Riojano Integral (Cori), La Rioja
  - Clínica Viedma, Viedma
- Australia (8):
  - Flinders Medical Centre, Bedford Park
  - Austin Hospital, Heidelberg
  - Cabrini Medical Centre, Malvern
  - St John of God Hospital Murdoch, Murdoch
  - Sir Charles Gairdner Hospital, Nedlands
  - Westmead Hospital, Westmead
  - Southern Medical Day Care Centre, Wollongong
  - Princess Alexandra Hospital, Woolloongabba
- Belgium (5):
  - Cliniques Universitaires Saint Luc, Brussels
  - Grand Hopital De Charleroi Site Les Viviers, Charleroi
  - UZ Leuven, Leuven
  - Clinique Saint Pierre, Ottignies
  - Algemeen Ziekenhuis Delta, Roeselare
- Brazil (16):
  - Fundacao Pio XII, Barretos
  - Cetus Oncologia, Belo Horizonte
  - Ynova Pesquisa Clinica, Florianópolis
  - Oncosite - Centro de Pesquisa Clínica em Oncologia Ltda, Ijuí
  - Liga Norte Riograndense Contra O Cancer, Natal
  - UPCO Unidade de Pesquisa Clinica em Oncologia, Pelotas
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Uniao Brasileira de Educacao e Assistencia Hospital Sao Lucas da PUCRS, Porto Alegre
  - Ministerio da Saude Instituto Nacional do Cancer, Rio de Janeiro
  - Oncoclinicas Rio de Janeiro S A, Rio de Janeiro
  - Instituto D Or de Pesquisa e Ensino IDOR, Rio de Janeiro
  - Fundacao Faculdade de Medicina Instituto do Cancer do Estado de Sao Paulo, São Paulo
  - Fundacao Antonio Prudente A C Camargo Cancer Center, São Paulo
  - Núcleo de Pesquisa São Camilo, São Paulo
  - IOS - Instituto de Oncologia de Sorocaba Dr. Gilson Delgado, Sorocaba
  - Hospital Evangélico de Cachoeiro de Itapemirim, Vitória
- Canada (4):
  - William Osler Health System, Brampton, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - McGill University Health Centre, Montreal, Quebec
- China (32):
  - Beijing Friendship Hospital Capital Medical University, Beijing
  - Beijing Cancer Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - Beijing Chest hospital, Capital medical university, Beijing
  - Jilin cancer hospital, Changchun
  - Hunan Cancer hospital, Changsha
  - The First People's Hospital Of Changzhou, Changzhou
  - Sichuan Cancer Hospital, Chengdu
  - West China Hospital Sichuan University, Chengdu
  - Southwest Hospital, Chongqing
  - The First Affiliated Hospital Sun Yat sen University, Guangzhou
  - Sun Yat-Sen Memorial Hospital Sun Yat-sen University, Guangzhou
  - Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou
  - The Second Affiliated Hospital of Zhejiang University College of Medicine, Hangzhou
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin medical university cancer hospital, Harbin
  - Huizhou Municipal Central Hospital, Huizhou
  - Taizhou Hospital of Zhejiang Province, Linhai
  - Nantong Tumor Hospital, Nantong
  - Ruijin Hospital Shanghai Jiao Tong University, Shanghai
  - Shanghai Chest Hospital, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai East Hospital, Shanghai
  - Shengjing Hospital Of China Medical University, Shenyang
  - Tianjin Medical University General Hospital, Tianjin
  - Cancer Hospital of Xinjiang Medical University, Ürümqi
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - TongJi Hospital of TongJi Medical College of Huazhong University of Science & Technology, Wuhan
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an
  - Yantai Yuhuangding Hospital, Yantai
  - Henan Cancer Hospital, Zhengzhou
- France (13):
  - Institut Bergonie, Bordeaux
  - Hospices Civils de Lyon HCL, Bron
  - CHU de Grenoble Hopital Albert Michallon, La Tronche
  - Institute Coeur Poumon, Lille
  - CHU de Limoges, Limoges
  - Hopital Nord, Marseille
  - Institut Curie, Paris
  - Hopital Tenon, Paris
  - CHU Bordeaux, Pessac
  - CHU Nantes, Sain-Herblain
  - HIA Begin, Saint-Mandé
  - CHU Bretonneau, Tours
  - Institut Gustave Roussy, Villejuif
- Germany (11):
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Helios Klinikum Emil von Behring GmbH, Berlin
  - Kliniken der Stadt Koeln gGmbH, Cologne
  - Universitaetsklinikum Essen, Essen
  - Asklepios Klinik Gauting GmbH - Asklepios Fachkliniken Munchen-Gauting, Gauting
  - Städtisches Krankenhaus Martha-Maria Halle-Dölau gGmbH, Halle
  - Thoraxklinik am Universitatsklinikum Heidelberg, Heidelberg
  - Onkologische Schwerpunktpraxis, Heilbronn
  - POIS Leipzig GbR, Leipzig
  - Pius-Hospital Oldenburg, Oldenburg
  - Robert-Bosch-Krankenhaus - Klinik Schillerhoehe, Stuttgart
- Hungary (6):
  - Orszagos Koranyi Tbc es Pulmonologiai Intezet, Budapest
  - Veszprém Megyei Tudőgyógyintézet, Farkasgyepü
  - Mátrai Gyógyintézet-Bronchológia, Gyöngyös
  - Fejer Varmegyei Szent Gyorgy Egyetemi Oktatokorhaz, Székesfehérvár
  - Markusovszky Egyetemi Oktatokorhaz, Szombathely
  - Tudogyogyintezet Torokbalint, Törökbálint
- India (5):
  - Basavatarakam Indo-American Hospital, Hyderabad
  - Tata Medical Center, Kolkata
  - Tata Memorial Hospital, Mumbai
  - HCG Manavta Cancer Centre, Nashik
  - Noble Hospital Pvt Ltd, Pune
- Israel (6):
  - Rambam Health Corporation, Haifa
  - Hadassah Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (13):
  - Ospedale San Giuseppe Moscati di Avellino, Avellino
  - Azienda Ospedaliero Univ. Policlinico Gaspare Rodolico, Catania
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Europeo di Oncologia, Milan
  - San Gerardo Hospital, Monza
  - Ospedale Monaldi, Napoli
  - Aou San Luigi Gonzaga, Orbassano
  - Ospedale S. Maria Delle Croci, Ravenna
  - Irccs Gemelli, Roma
  - Istituto Clinico Humanitas, Rozzano
- Japan (20):
  - Juntendo University Hospital, Bunkyō City
  - National Cancer Center Hospital, Chūōku
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - National Hospital Organization Himeji Medical Center, Himeji
  - Kansai Medical University Hospital, Hirakata
  - Kanazawa University Hospital, Kanazawa
  - National Cancer Center Hospital East, Kashiwa
  - Kurume University Hospital, Kurume
  - Matsusaka Municipal Hospital, Matsusaka
  - Niigata Cancer Center Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Kindai University Hospital, Osaka Sayama Shi
  - National Hospital Organization Shibukawa Medical Center, Shibukawa
  - The Cancer Institute Hospital of JFCR, Tokyo
  - National Hospital Organization Tokyo Medical Center, Tokyo
  - Ehime University Hospital, Toon-shi
  - National Hospital Organization Osaka Toneyama Medical Center, Toyonaka-shi
  - Wakayama Medical University Hospital, Wakayama
  - National Hospital Organization Iwakuni Clinical Center, Yamaguchi
  - National Hospital Organization Yamaguchi Ube Medical Center, Yamaguchi
- Malaysia (6):
  - Hospital Pulau Pinang, George Town
  - Hospital Sultan Ismail, Johor Bahru
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan
  - Beacon Hospital Sdn Bhd, Petaling Jaya
- Mexico (8):
  - Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara
  - CIMOVA, Morals Vargas Centro de Investigación SC, León
  - Mexico Centre for Clinical Research, S.A. de C.V., Mexico City
  - Médica Sur, Mexico City
  - Health Pharma Professional Research, México
  - Instituto Nacional de Cancerologia, México
  - i Can Oncology Center, Monterrey
  - Oncologia Integral Satelite, Naucalpan
- Netherlands (4):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Rijnstate Ziekenhuis, Arnhem
  - Ziekenhuis St Jansdal, Harderwijk
  - UMC Radboud, Nijmegen
- Poland (6):
  - Centrum Onkologii im Prof F Lukaszczyka, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Szpitale Pomorskie Sp z o o, Gdynia
  - Warminsko-Mazurskie Centrum Chorob Pluc w Olsztynie, Olsztyn
  - Private Specialist Hospitals - MedPolonia, Poznan
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut Badawczy, Warsaw
- Portugal (4):
  - Uls Santa Maria - Hosp. Pulido Valente, Lisbon
  - Uls Santo Antonio - Hosp. Santo Antonio, Porto
  - Hosp. Cuf Porto, Porto
  - Instituto Portugues de Oncologia, Porto
- Pan American Center for Oncology Trials LLC, Rio Piedras, Puerto Rico
- Russia (15):
  - Irkutsk Regional Oncology Dispensary, Irkutsk
  - Moscow City Oncology Hospital № 62, Krasnogorsk
  - Krasnoyarsk Regional Oncology Dispensary, Krasnoyarsk
  - Leningrad Regional Oncology Dispensary, Kuzmolovsky
  - MCK, Moscow
  - City Clinical Hospital #1, Nal'chik
  - Nizhny Novgorod Regional Oncological Dispensary, Nizhny Novgorod
  - Omsk Clinical Oncology Dispensary, Omsk
  - Current medical technologies, Saint Petersburg
  - Oncology Medical Clinics AV Medical group, Saint Petersburg
  - N.N. Petrov Research Institute Of Oncology, Saint Petersburg
  - Tambov Regional Oncology Clinical Dispansary, Tambov
  - Tomsk Cancer Research Institute, Tomsk
  - Bashkir State Medical University, Ufa
  - Yaroslavl Regional Clinical Oncology Hospital, Yaroslavl
- South Korea (9):
  - Inje University Haeundae Paik Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Seoul National University Bundang Hospital, Seongnam-si
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Mary s Hospital, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (16):
  - Hosp Univ A Coruna, A Coruña
  - Inst. Cat. D'Oncologia-Badalona, Badalona
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hosp. Univ. Quiron Dexeus, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Univ. de Burgos, Burgos
  - Institut Català D'Oncologia Girona, Girona
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hosp. Univ. Pta. de Hierro Majadahonda, Majadahonda
  - Hosp Regional Univ de Malaga, Málaga
  - Clinica Univ. de Navarra, Pamplona
  - Hosp. Virgen Del Rocio, Seville
  - Hosp. Gral. Univ. Valencia, Valencia
  - Hosp. Clinico Univ. Lozano Blesa, Zaragoza
- Taiwan (8):
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - E-DA Hospital, Kaohsiung City
  - Chang Gung Medical Foundation, Kaohsiung City
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- Thailand (4):
  - Phramongkutklao Hospital and Medical College, Bangkok
  - Siriraj Hospital, Bangkok
  - Chiang Mai University, Chiang Mai
  - Songklanagarind Hospital, Prince of Songkla University, Songkhla
- Turkey (Türkiye) (10):
  - Adana City Hospital, Adana
  - Başkent University Medical Faculty Adana Application and Research Center, Adana
  - Gazi University Hospital, Ankara
  - Ankara Bilkent City Hospital, Ankara
  - Trakya University Medical Faculty, Edirne
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi Ic Hastaliklari Anabilim Dali Medikal Onkoloji Bd, Istanbul
  - Medipol Mega University Hospital, Istanbul
  - T C Saglik Bakanlıgi Goztepe Prof Dr Suleyman Yalcın Sehir Hastanesi, Istanbul
  - Medical Point, Izmir
  - Necmettin Erbakan University Meram Medical Faculty, Konya
- Ukraine (5):
  - Dnipropetrovsk State Medical Academy, Dnipropetrovsk City Multifield Clinical Hospital # 4, Dnipro
  - Municipal non-profit enterprise 'Regional Center of Oncology', Kharkiv
  - Medical Center 'Ok Clinic' of LLC 'International Institute of Clinical Studies', Kyiv
  - National Cancer Institute, Kyiv
  - Municipal Oncology Centre of Uzhgorod Central Municipal Clinical Hospitlal, Uzhhorod
- United Kingdom (7):
  - Edinburgh Cancer Centre Western General, Edinburgh
  - UCL Cancer Institute, London
  - Chelsea And Westminster Hospital, London
  - The Royal Marsden NHS Trust, London
  - Christie NHS Foundation Trust, Manchester
  - Nottingham University Hospitals NHS Trust, Nottingham
  - The Royal Marsden NHS Trust, Sutton

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency

REFERENCES:
- [Derived] Yang JC, Lu S, Hayashi H, Felip E, Spira AI, Girard N, Kim YJ, Lee SH, Ostapenko Y, Danchaivijitr P, Liu B, Alip A, Korbenfeld E, Mourao Dias J, Besse B, Passaro A, Lee KH, Xiong H, How SH, Cheng Y, Chang GC, Yoshioka H, Thomas M, Nguyen D, Ou SI, Mukhedkar S, Prabhash K, D'Arcangelo M, Alatorre-Alexander J, Vazquez Limon JC, Alves S, Stroyakovskiy D, Peregudova M, Sendur MAN, Yazici O, Califano R, Gutierrez Calderon V, de Marinis F, Kim SW, Gadgeel SM, Owen S, Xie J, Sun T, Mehta J, Venkatasubramanian R, Ennis M, Fennema E, Daksh M, Roshak A, Man J, Knoblauch RE, Bauml JM, Baig M, Shah S, Sethi S, Cho BC; MARIPOSA Investigators. Overall Survival with Amivantamab-Lazertinib in EGFR-Mutated Advanced NSCLC. N Engl J Med. 2025 Oct 30;393(17):1681-1693. doi: 10.1056/NEJMoa2503001. Epub 2025 Sep 7. PMID 40923797
- [Derived] Cho BC, Lu S, Felip E, Spira AI, Girard N, Lee JS, Lee SH, Ostapenko Y, Danchaivijitr P, Liu B, Alip A, Korbenfeld E, Mourao Dias J, Besse B, Lee KH, Xiong H, How SH, Cheng Y, Chang GC, Yoshioka H, Yang JC, Thomas M, Nguyen D, Ou SI, Mukhedkar S, Prabhash K, D'Arcangelo M, Alatorre-Alexander J, Vazquez Limon JC, Alves S, Stroyakovskiy D, Peregudova M, Sendur MAN, Yazici O, Califano R, Gutierrez Calderon V, de Marinis F, Passaro A, Kim SW, Gadgeel SM, Xie J, Sun T, Martinez M, Ennis M, Fennema E, Daksh M, Millington D, Leconte I, Iwasawa R, Lorenzini P, Baig M, Shah S, Bauml JM, Shreeve SM, Sethi S, Knoblauch RE, Hayashi H; MARIPOSA Investigators. Amivantamab plus Lazertinib in Previously Untreated EGFR-Mutated Advanced NSCLC. N Engl J Med. 2024 Oct 24;391(16):1486-1498. doi: 10.1056/NEJMoa2403614. Epub 2024 Jun 26. PMID 38924756
- [Derived] Cho BC, Felip E, Hayashi H, Thomas M, Lu S, Besse B, Sun T, Martinez M, Sethi SN, Shreeve SM, Spira AI. MARIPOSA: phase 3 study of first-line amivantamab + lazertinib versus osimertinib in EGFR-mutant non-small-cell lung cancer. Future Oncol. 2022 Feb;18(6):639-647. doi: 10.2217/fon-2021-0923. Epub 2021 Dec 16. PMID 34911336

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Currently, results posted till cut-off date 11-Aug-2023 (primary completion date). After analyzing primary analysis of progression free survival, participants were transitioned to an open-label extension (OLE) phase. Participants who continue to benefit from study treatment(s), as determined by investigator, may continue to receive access to study treatment(s) within study by transferring to long-term extension phase. OLE phase is still ongoing and results will be posted upon study completion.
Groups:
- Experimental: Arm A (Open-label): Amivantamab + Lazertinib: Participants received combination therapy of amivantamab 1050 milligrams (mg) for body weight (BW) less than (<) 80 kilograms (kg) or 1400 mg for BW greater than or equal to (>=) 80 kg intravenous (IV) infusion once weekly in 28-day treatment cycles: at Cycle 1 Days 1/2 (split dose, Day 1: 350 mg regardless of BW; Day 2: 700 mg or 1050 mg [if BW >=80 kg]), 8, 15, and 22 and then once every 2 weeks (at Day 1 and 15) from Cycle 2 onwards; and lazertinib 240 mg (3 tablets of 80 mg) orally once daily. Participants continued treatment until disease progression, participant consent withdrawal, adverse event, investigator's decision, or initiation of new systemic anti-cancer treatment.
- Active Comparator: Arm B (Double-blind): Osimertinib+Placebo Matching Lazertinib: Participants received osimertinib 80 mg capsule orally once daily along with 3 tablets of matching placebo of lazertinib 240 mg tablets orally once daily from Cycle 1 Day 1 until disease progression, participant consent withdrawal, adverse event, investigator's decision, or initiation of new systemic anti-cancer treatment.
- Experimental: Arm C (Double-blind): Lazertinib+Placebo Matching Osimertinib: Participants received lazertinib 240 mg (3 tablets of 80 mg) orally once daily along with single capsule of matching placebo of osimertinib 80 mg orally once daily from Cycle 1 Day 1 until disease progression, participant consent withdrawal, adverse event, investigator's decision, or initiation of new systemic anti-cancer treatment.
Period: Overall Study
Arm/Group | Experimental: Arm A (Open-label): Amivantamab + Lazertinib | Active Comparator: Arm B (Double-blind): Osimertinib+Placebo Matching Lazertinib | Experimental: Arm C (Double-blind): Lazertinib+Placebo Matching Osimertinib
Started | 429 | 429 | 216
Treated | 421 | 428 | 213
Completed | 94 | 113 | 54
Not Completed | 335 | 316 | 162
Not completed — Withdrawal by Subject | 19 | 18 | 13
Not completed — Lost to Follow-up | 3 | 1 | 0
Not completed — Ongoing | 313 | 297 | 149

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Arm A (Open-label): Amivantamab + Lazertinib | Active Comparator: Arm B (Double-blind): Osimertinib+Placebo Matching Lazertinib | Experimental: Arm C (Double-blind): Lazertinib+Placebo Matching Osimertinib | Total
Number analyzed (Participants) | 429 | 429 | 216 | 1074
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (10.63) | 61.9 (11.52) | 61.3 (10.69) | 62.1 (11.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 275 | 251 | 136 | 662
  Male | 154 | 178 | 80 | 412
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 56 | 45 | 24 | 125
  Not Hispanic or Latino | 371 | 382 | 190 | 943
  Unknown or Not Reported | 2 | 2 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 7 | 4 | 18
  Asian | 250 | 251 | 128 | 629
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 2
  Black or African American | 4 | 3 | 4 | 11
  White | 164 | 165 | 79 | 408
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 2 | 1 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 8 | 11 | 6 | 25
  AUSTRALIA | 5 | 7 | 1 | 13
  BELGIUM | 2 | 4 | 1 | 7
  BRAZIL | 38 | 22 | 9 | 69
  CANADA | 0 | 0 | 2 | 2
  CHINA | 81 | 79 | 43 | 203
  FRANCE | 12 | 11 | 6 | 29
  GERMANY | 2 | 5 | 2 | 9
  HUNGARY | 2 | 0 | 1 | 3
  INDIA | 6 | 16 | 3 | 25
  ISRAEL | 3 | 3 | 2 | 8
  ITALY | 11 | 8 | 5 | 24
  JAPAN | 29 | 32 | 17 | 78
  MALAYSIA | 27 | 23 | 10 | 60
  MEXICO | 12 | 14 | 5 | 31
  NETHERLANDS | 1 | 2 | 0 | 3
  POLAND | 7 | 6 | 0 | 13
  PORTUGAL | 4 | 2 | 2 | 8
  RUSSIAN FEDERATION | 17 | 15 | 8 | 40
  SOUTH KOREA | 63 | 68 | 33 | 164
  SPAIN | 26 | 33 | 15 | 74
  TAIWAN | 24 | 15 | 13 | 52
  THAILAND | 15 | 9 | 5 | 29
  TURKEY | 15 | 21 | 4 | 40
  UKRAINE | 10 | 11 | 10 | 31
  UNITED KINGDOM | 2 | 7 | 2 | 11
  UNITED STATES | 7 | 5 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 as Assessed by Blinded Independent Central Review (BICR)
Description: PFS was defined as the time from randomization until the date of objective disease progression based on BICR using RECIST version 1.1 or death (by any cause) the absence of progression, whichever came first. Disease progression was defined using RECIST 1.1 as a 20 percent (%) increase in the sum of diameters of target measurable lesions above the smallest sum observed, with a minimum absolute increase of 5 millimeters (mL). Participants who have not progressed or have not died at the time of analysis were censored at the time of the latest date of their last evaluable RECIST version 1.1 assessment.
Time Frame: From randomization to either disease progression or death whichever occurs first (up to 32.8 months)
Population: Full analysis set (FAS) included all randomized participants, classified according to their assigned treatment arm regardless of the actual treatment received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Experimental: Arm A (Open-label): Amivantamab + Lazertinib | Active Comparator: Arm B (Double-blind): Osimertinib+Placebo Matching Lazertinib | Experimental: Arm C (Double-blind): Lazertinib+Placebo Matching Osimertinib
Number analyzed (Participants) | 429 | 429 | 216
Months | 23.72 [19.12 to 27.66] | 16.59 [14.78 to 18.46] | 18.46 [14.75 to 20.11]
Statistical Analysis 1: Comparison: Experimental: Arm A (Open-label): Amivantamab + Lazertinib vs Active Comparator: Arm B (Double-blind): Osimertinib+Placebo Matching Lazertinib; Test type: Superiority; p = 0.0002, Log Rank; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.58 to 0.85] — HR and its 95% CI was estimated based on a stratified Cox's regression model with treatment as the sole explanatory variable

2. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival is defined as the time from the date of randomization to the date of participant's death due to any cause.
Time Frame: Approximately 60 months (time from the date of randomization until the date of death due to any cause)
Reporting Status: Not Posted, anticipated posting 2028-06

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants who achieve either a complete response (CR) or partial response (PR) as defined by BICR using RECIST v1.1 criteria.
Time Frame: Approximately 32.8 months
Reporting Status: Not Posted, anticipated posting 2028-06

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from the date of first documented response (CR or PR) until the date of documented progression or death, whichever comes first, only for participants who achieve CR or PR as determined by the investigator using RECIST v1.1 criteria.
Time Frame: Approximately 32.8 months
Reporting Status: Not Posted, anticipated posting 2028-06

5. Secondary Outcome: Progression-Free Survival After First Subsequent Therapy (PFS2)
Description: The PFS2 is defined as the time from randomization until the date of second objective disease progression, after initiation of subsequent anticancer therapy, based on investigator assessment (after that used for PFS) or death, whichever comes first.
Time Frame: Approximately 60 months
Reporting Status: Not Posted, anticipated posting 2028-06

6. Secondary Outcome: Time to Symptomatic Progression (TTSP)
Description: TTSP is defined as the time from randomization to documentation in the electronic case report form (eCRF) of any of the following (whichever occurs earlier): onset of new symptoms or symptom worsening that is considered by the investigator to be related to lung cancer and requires either a change in anticancer treatment and/or clinical intervention to manage symptoms.
Time Frame: Approximately 60 months
Reporting Status: Not Posted, anticipated posting 2028-06

7. Secondary Outcome: Intracranial PFS
Description: Intracranial PFS is defined as the time from randomization until the date of objective intracranial disease progression or death, whichever comes first, based on BICR using RECIST v1.1.
Time Frame: Approximately 60 months
Reporting Status: Not Posted, anticipated posting 2028-06

8. Secondary Outcome: Incidence and Severity of Adverse Events (AEs)
Description: Incidence and severity of treatment emergent adverse events (TEAEs) will be reported. Any adverse event occurring at or after the initial administration of study treatment through the day of last dose plus 30 days, or until the start of subsequent anticancer therapy (if earlier), is considered to be treatment emergent.
Time Frame: Approximately 60 months
Reporting Status: Not Posted, anticipated posting 2028-06

9. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities
Description: Number of participants with clinical laboratory abnormalities (serum chemistry, hematology, blood coagulation, and urine samples) will be reported.
Time Frame: Approximately 60 months
Reporting Status: Not Posted, anticipated posting 2028-06

10. Secondary Outcome: Number of Participants With Vital Signs Abnormalities
Description: Number of participants with vital signs abnormalities (temperature, heart rate, respiratory rate, oxygen saturation, blood pressure) will be reported.
Time Frame: Approximately 60 months
Reporting Status: Not Posted, anticipated posting 2028-06

11. Secondary Outcome: Number of Participants With Physical Examination Abnormalities
Description: Number of participants with physical examination abnormalities will be reported.
Time Frame: Approximately 60 months
Reporting Status: Not Posted, anticipated posting 2028-06

12. Secondary Outcome: Serum Concentration of Amivantamab
Description: Serum samples will be analyzed to determine concentrations of Amivantamab.
Time Frame: Approximately 60 months
Reporting Status: Not Posted, anticipated posting 2028-06

13. Secondary Outcome: Plasma Concentration of Lazertinib
Description: Plasma samples will be analyzed to determine concentrations of Lazertinib.
Time Frame: Approximately 60 months
Reporting Status: Not Posted, anticipated posting 2028-06

14. Secondary Outcome: Number of Participants With Anti-Amivantamab Antibodies
Description: Number of participants with antibodies to amivantamab will be reported.
Time Frame: Approximately 60 months
Reporting Status: Not Posted, anticipated posting 2028-06

15. Secondary Outcome: Change From Baseline in Non-Small Cell Lung Cancer - Symptom Assessment Questionnaire (NCSLC-SAQ)
Description: The NSCLC-SAQ contains 7 items that assess cough, pain, dyspnea, fatigue, and poor appetite over a 7-day recall period. Each multi-item scale and individual item will be summarized using count and percent by visit.
Time Frame: Baseline up to approximately 60 months
Reporting Status: Not Posted, anticipated posting 2028-06

16. Secondary Outcome: Change From Baseline in European Organization of Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC-QLQ-C30)
Description: EORTC-QLQ-C30 is a core 30-item questionnaire for evaluating the health-related quality of life (HRQoL) of participants participating in cancer clinical studies.
Time Frame: Baseline up to approximately 60 months
Reporting Status: Not Posted, anticipated posting 2028-06

ADVERSE EVENTS:
Time Frame: From baseline (Day 1 of Cycle 1) up to 32.8 months
Description: The safety set included randomized participants who received at least 1 dose of study treatment.
Arm/Group | Experimental: Arm A (Open-label): Amivantamab + Lazertinib | Active Comparator: Arm B (Double-blind): Osimertinib+Placebo Matching Lazertinib | Experimental: Arm C (Double-blind): Lazertinib+Placebo Matching Osimertinib
All-Cause Mortality (participants affected / at risk) | 96/421 | 116/428 | 56/213
Serious Adverse Events (participants affected / at risk) | 205/421 | 143/428 | 75/213
Other Adverse Events (participants affected / at risk) | 419/421 | 409/428 | 210/213
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Arm A (Open-label): Amivantamab + Lazertinib (N=421) | Active Comparator: Arm B (Double-blind): Osimertinib+Placebo Matching Lazertinib (N=428) | Experimental: Arm C (Double-blind): Lazertinib+Placebo Matching Osimertinib (N=213)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 26 | 10 | 8
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 9 | 17 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 | 8 | 3
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 11 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypersensitivity Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 17 | 21 | 7
Covid-19 (Infections and infestations) | 10 | 10 | 3
Cellulitis (Infections and infestations) | 4 | 0 | 2
Sepsis (Infections and infestations) | 3 | 1 | 0
Septic Shock (Infections and infestations) | 3 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 3 | 1 | 1
Dermatitis Infected (Infections and infestations) | 2 | 0 | 0
Achromobacter Infection (Infections and infestations) | 1 | 0 | 0
Acinetobacter Sepsis (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 1 | 0
Appendicitis Perforated (Infections and infestations) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Covid-19 Pneumonia (Infections and infestations) | 1 | 1 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Device Related Infection (Infections and infestations) | 1 | 0 | 0
Gastrointestinal Infection (Infections and infestations) | 1 | 0 | 0
Pneumonia Aspiration (Infections and infestations) | 1 | 1 | 0
Post Procedural Infection (Infections and infestations) | 1 | 0 | 0
Pustule (Infections and infestations) | 1 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 2
Skin Infection (Infections and infestations) | 1 | 0 | 0
Staphylococcal Sepsis (Infections and infestations) | 1 | 0 | 0
Subcutaneous Abscess (Infections and infestations) | 1 | 0 | 0
Tinea Cruris (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 1 | 0
Wound Infection (Infections and infestations) | 1 | 0 | 0
Arthritis Bacterial (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1
Dengue Fever (Infections and infestations) | 0 | 0 | 1
Epididymitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 0
Herpes Virus Infection (Infections and infestations) | 0 | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0
Otitis Media Chronic (Infections and infestations) | 0 | 0 | 1
Periodontitis (Infections and infestations) | 0 | 0 | 1
Scrub Typhus (Infections and infestations) | 0 | 1 | 0
Soft Tissue Infection (Infections and infestations) | 0 | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1
Infusion Related Reaction (Injury, poisoning and procedural complications) | 9 | 0 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 4 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 3 | 0 | 0
Accidental Overdose (Injury, poisoning and procedural complications) | 1 | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Muscle Rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radiation Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Recall Phenomenon (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 2 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head Injury (Injury, poisoning and procedural complications) | 0 | 2 | 0
Procedural Pneumothorax (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radiation Pneumonitis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 12 | 2 | 1
Venous Thrombosis (Vascular disorders) | 4 | 0 | 0
Venous Thrombosis Limb (Vascular disorders) | 4 | 0 | 3
Jugular Vein Thrombosis (Vascular disorders) | 2 | 0 | 0
Circulatory Collapse (Vascular disorders) | 1 | 0 | 0
Embolism Venous (Vascular disorders) | 1 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 1 | 0 | 0
Peripheral Artery Thrombosis (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0
Embolism (Vascular disorders) | 0 | 2 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 | 1 | 0
Superior Vena Cava Syndrome (Vascular disorders) | 0 | 1 | 0
Sudden Death (General disorders) | 4 | 1 | 1
Asthenia (General disorders) | 3 | 1 | 1
Death (General disorders) | 3 | 2 | 1
Fatigue (General disorders) | 2 | 2 | 1
General Physical Health Deterioration (General disorders) | 2 | 0 | 0
Oedema Peripheral (General disorders) | 2 | 0 | 0
Pyrexia (General disorders) | 2 | 1 | 0
Generalised Oedema (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 1 | 1 | 0
Mucosal Inflammation (General disorders) | 1 | 0 | 0
Oedema (General disorders) | 1 | 0 | 0
Peripheral Swelling (General disorders) | 1 | 0 | 0
Chest Pain (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 2 | 1
Colitis (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Gastric Ulcer Perforation (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Ileus Paralytic (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 1 | 0 | 0
Mallory-Weiss Syndrome (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0 | 0
Peptic Ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1 | 0
Intra-Abdominal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Mesenteric Vascular Occlusion (Gastrointestinal disorders) | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 4 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Failure to Thrive (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 4 | 0 | 0
Pericardial Effusion (Cardiac disorders) | 4 | 5 | 4
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0 | 0
Arteriosclerosis Coronary Artery (Cardiac disorders) | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 1 | 0
Atrioventricular Block Second Degree (Cardiac disorders) | 1 | 0 | 0
Cardiac Failure (Cardiac disorders) | 1 | 5 | 1
Cardiac Tamponade (Cardiac disorders) | 1 | 0 | 0
Cardiopulmonary Failure (Cardiac disorders) | 1 | 0 | 0
Cardiovascular Insufficiency (Cardiac disorders) | 1 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 1 | 0 | 0
Myocardial Rupture (Cardiac disorders) | 1 | 0 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 2 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 2
Myocardial Injury (Cardiac disorders) | 0 | 0 | 1
Cerebral Infarction (Nervous system disorders) | 2 | 4 | 1
Cerebellar Ataxia (Nervous system disorders) | 1 | 0 | 0
Cerebral Haemorrhage (Nervous system disorders) | 1 | 1 | 0
Cerebral Thrombosis (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 2 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1
Haemorrhagic Stroke (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0
Ischaemic Cerebral Infarction (Nervous system disorders) | 1 | 0 | 0
Loss of Consciousness (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 1 | 1
Superior Sagittal Sinus Thrombosis (Nervous system disorders) | 1 | 0 | 0
Brain Oedema (Nervous system disorders) | 0 | 2 | 0
Cognitive Disorder (Nervous system disorders) | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 2 | 0
Facial Paralysis (Nervous system disorders) | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 1
Intracranial Pressure Increased (Nervous system disorders) | 0 | 0 | 1
Meningism (Nervous system disorders) | 0 | 1 | 0
Paraparesis (Nervous system disorders) | 0 | 1 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 0 | 1
Spinal Cord Compression (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 8 | 6 | 4
Eastern Cooperative Oncology Group Performance Status Worsened (Investigations) | 2 | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 1 | 4 | 4
Troponin I Increased (Investigations) | 1 | 0 | 0
Blood Bilirubin Increased (Investigations) | 0 | 1 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 1 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 1 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 7 | 0 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Drug Eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Chronic Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
High-Grade B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ureteral Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 1
Bone Marrow Failure (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 2 | 0 | 0
Renal Impairment (Renal and urinary disorders) | 1 | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 2 | 1
Chronic Kidney Disease (Renal and urinary disorders) | 0 | 1 | 0
Renal Colic (Renal and urinary disorders) | 0 | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 1 | 1
Urogenital Disorder (Renal and urinary disorders) | 0 | 1 | 0
Giant Papillary Conjunctivitis (Eye disorders) | 1 | 0 | 0
Keratitis (Eye disorders) | 1 | 0 | 0
Papilloedema (Eye disorders) | 1 | 0 | 0
Optic Atrophy (Eye disorders) | 0 | 0 | 1
Optic Ischaemic Neuropathy (Eye disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 1
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1
Device Dislocation (Product Issues) | 2 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 1
Mental Status Changes (Psychiatric disorders) | 1 | 0 | 0
Confusional State (Psychiatric disorders) | 0 | 0 | 1
Major Depression (Psychiatric disorders) | 0 | 0 | 1
Panic Disorder (Psychiatric disorders) | 0 | 1 | 0
Genital Tract Inflammation (Reproductive system and breast disorders) | 1 | 0 | 0
Pelvic Pain (Reproductive system and breast disorders) | 1 | 0 | 0
Pleurodesis (Surgical and medical procedures) | 1 | 0 | 0
Cholecystectomy (Surgical and medical procedures) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Arm A (Open-label): Amivantamab + Lazertinib (N=421) | Active Comparator: Arm B (Double-blind): Osimertinib+Placebo Matching Lazertinib (N=428) | Experimental: Arm C (Double-blind): Lazertinib+Placebo Matching Osimertinib (N=213)
Rash (Skin and subcutaneous tissue disorders) | 260 | 131 | 95
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 122 | 55 | 45
Pruritus (Skin and subcutaneous tissue disorders) | 99 | 73 | 36
Dry Skin (Skin and subcutaneous tissue disorders) | 67 | 60 | 38
Skin Fissures (Skin and subcutaneous tissue disorders) | 40 | 23 | 5
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 27 | 8 | 8
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 24 | 15 | 13
Skin Ulcer (Skin and subcutaneous tissue disorders) | 22 | 2 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 15 | 20 | 27
Paronychia (Infections and infestations) | 288 | 121 | 61
Covid-19 (Infections and infestations) | 104 | 97 | 39
Conjunctivitis (Infections and infestations) | 46 | 7 | 7
Upper Respiratory Tract Infection (Infections and infestations) | 37 | 44 | 13
Urinary Tract Infection (Infections and infestations) | 30 | 20 | 10
Folliculitis (Infections and infestations) | 27 | 7 | 9
Pneumonia (Infections and infestations) | 22 | 22 | 11
Diarrhoea (Gastrointestinal disorders) | 123 | 189 | 68
Constipation (Gastrointestinal disorders) | 122 | 55 | 36
Stomatitis (Gastrointestinal disorders) | 122 | 90 | 38
Nausea (Gastrointestinal disorders) | 90 | 58 | 38
Vomiting (Gastrointestinal disorders) | 52 | 23 | 23
Haemorrhoids (Gastrointestinal disorders) | 41 | 9 | 8
Dyspepsia (Gastrointestinal disorders) | 32 | 18 | 9
Abdominal Pain Upper (Gastrointestinal disorders) | 26 | 18 | 9
Hypoalbuminaemia (Metabolism and nutrition disorders) | 204 | 26 | 17
Decreased Appetite (Metabolism and nutrition disorders) | 101 | 76 | 31
Hypocalcaemia (Metabolism and nutrition disorders) | 87 | 35 | 15
Hypokalaemia (Metabolism and nutrition disorders) | 60 | 30 | 12
Hyponatraemia (Metabolism and nutrition disorders) | 38 | 37 | 22
Hyperglycaemia (Metabolism and nutrition disorders) | 26 | 20 | 5
Oedema Peripheral (General disorders) | 150 | 24 | 24
Asthenia (General disorders) | 77 | 46 | 31
Fatigue (General disorders) | 68 | 41 | 22
Pyrexia (General disorders) | 49 | 36 | 20
Mucosal Inflammation (General disorders) | 44 | 12 | 8
Peripheral Swelling (General disorders) | 22 | 5 | 2
Chest Pain (General disorders) | 18 | 20 | 11
Non-Cardiac Chest Pain (General disorders) | 13 | 18 | 11
Infusion Related Reaction (Injury, poisoning and procedural complications) | 261 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 152 | 55 | 47
Aspartate Aminotransferase Increased (Investigations) | 121 | 58 | 43
Gamma-Glutamyltransferase Increased (Investigations) | 61 | 31 | 19
Blood Alkaline Phosphatase Increased (Investigations) | 52 | 22 | 16
Blood Lactate Dehydrogenase Increased (Investigations) | 49 | 24 | 21
Weight Decreased (Investigations) | 37 | 37 | 5
Blood Creatinine Increased (Investigations) | 31 | 49 | 27
Blood Creatine Phosphokinase Increased (Investigations) | 14 | 19 | 16
Weight Increased (Investigations) | 12 | 9 | 12
Paraesthesia (Nervous system disorders) | 58 | 25 | 33
Headache (Nervous system disorders) | 55 | 54 | 38
Dizziness (Nervous system disorders) | 49 | 31 | 13
Neuropathy Peripheral (Nervous system disorders) | 41 | 3 | 23
Hypoaesthesia (Nervous system disorders) | 28 | 7 | 18
Peripheral Sensory Neuropathy (Nervous system disorders) | 23 | 10 | 19
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 70 | 32 | 50
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 64 | 22 | 21
Myalgia (Musculoskeletal and connective tissue disorders) | 52 | 19 | 11
Back Pain (Musculoskeletal and connective tissue disorders) | 48 | 45 | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 38 | 59 | 25
Cough (Respiratory, thoracic and mediastinal disorders) | 65 | 88 | 37
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 63 | 16 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 49 | 62 | 25
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 33 | 14 | 5
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 22 | 19 | 14
Anaemia (Blood and lymphatic system disorders) | 96 | 91 | 42
Thrombocytopenia (Blood and lymphatic system disorders) | 66 | 84 | 20
Leukopenia (Blood and lymphatic system disorders) | 26 | 66 | 15
Lymphopenia (Blood and lymphatic system disorders) | 22 | 31 | 15
Neutropenia (Blood and lymphatic system disorders) | 20 | 56 | 7
Deep Vein Thrombosis (Vascular disorders) | 56 | 10 | 6
Hypotension (Vascular disorders) | 29 | 4 | 2
Hypertension (Vascular disorders) | 21 | 17 | 12
Insomnia (Psychiatric disorders) | 41 | 48 | 13
Dry Eye (Eye disorders) | 37 | 18 | 7
Hyperbilirubinaemia (Hepatobiliary disorders) | 28 | 14 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2023-11-14): https://cdn.clinicaltrials.gov/large-docs/80/NCT04487080/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT04487080/SAP_001.pdf